CLINICAL TRIAL: NCT03268915
Title: Assessment of the Reproducibility of the 3 Minutes Sit-to-stand Test in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Idiopathic Pulmonary Fibrosis (IPF) and the 3 Minutes Sit-to-stand Test
Acronym: ST2-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EssaisCliniques_TCL3-FPI
Record Dates: First submitted 2017-07-21; First posted 2017-08-31 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; 3 minutes sit-to-stand test; Interindividual reproductibility
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Walk Test

STUDY DESIGN:
Intervention Model Description: The investigators want to test the reproductibility of a 3 minutes sit-to-stand test in patients with idiopathic pulmonary fibrosis.
  For this, patient perform the test during 2 visits and the investigators are going to compare the results of the two visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with idiopathic pulmonary fibrosis (Experimental)
  Interventions: Diagnostic Test: 3 minutes sit-to-stand test

INTERVENTIONS:
Diagnostic Test: 3 minutes sit-to-stand test — 3 minutes sit-to-stand test, 1 minute sit-to-stand test, 6 minutes walk test will be performed 2 times for each patients 3 minutes sit-to-stand test with oxygen uptake measurement will be performed one time for each patient
  Other Names: 6 minutes walk test; 1 minute sit-to-stand test; 3 minutes sit-to-stand test with oxygen uptake measurement

SUMMARY:
This study is designed to evaluate the reproductibility and the performance of the 3 minutes sit-to-stand test in patients with idiopathic pulmonary fibrosis.

To do this, the investigators are recruiting 40 patients with idiopathic pulmonary fibrosis in 2 centers (Grenoble university hospital and Lyon university hospital).

Patients had to achieve an effort test on a cycle ergometer. 2 visits are planned in the hospital. During each visit, patients will perform a 3 minutes sit-to-stand test, a 1 minute sit-to-stand test and a 6 minutes walk test. During the second visit, patients will also perform a 3 minutes sit-to-stand test with measurement of oxygen uptake.

The investigators will then analyse the results by comparing numbers of cycle, functional response and symptoms during the 3 minutes sit-to-stand test of the 2 visits. The investigators will also compare the functional response obtained during the 3 minutes sit-to-stand test, the 1 minute sit-to-stand test and the 6 minutes walk test.

Finally, the investigators will compare the maximal values of oxygen uptake, respiration rate and expired volume obtained during the 3 minutes sit-to-stand test to the effort test on cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged less than 85 years
* patients with Idiopathic Pulmonary Fibrosis without any acute exacerbation during 4 months before the inclusion
* Non-opposition to participation in research
* Patient with 6 minutes walk test > 200 meters (with or without oxygen therapy)

Exclusion Criteria:

* Patient with reduced locomotor activity, or joint pain that compromises the performance of the tests
* Patient with 6 minutes walk test < 200 meters
* Patient with an other etiology of pulmonary fibrosis
* Other significant pulmonary diseases
* Patient with unstable cardiac disease
* Patient who may be, according to the investigator's assessment, not cooperating or respecting the obligations inherent in participating to the study.
* Opposition to participation in research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Reproductibility of the 3 minutes sit-to-stand test in patient with idiopathic pulmonary fibrosis | 2 days
  Evaluate the reproductibility for the number of rise and down during the 3 minutes sit-to-stand test of the 2 visits (the investigators will compare the number of rise and sit during the 3 minutes sit-to-stand test of the 2 visits to see if they are similar)

SECONDARY OUTCOMES:
Functional response during the 3 minutes sit-to-stand test: Oxygen saturation | 2 days
  Evaluate the reproductibility of functional response (oxygen saturation) during the 3 minutes sit-to-stand test
3 minutes sit-to-stand test compared to the 6 minutes walk test: oxygen saturation | 2 days
  compared oxygen saturation during the 3 minutes sit-to-stand test to the 6 minutes walk test
1 minute sit-to-stand test compared to 3 minutes sit-to-stand: oxygen saturation | 2 days
  Compared oxygen saturation during the 3 minutes sit-to-stand test with 1 minute sit-to-stand test
Functional response during the 3 minutes sit-to-stand test: Heart rate | 2 days
  Evaluate the reproductibility of functional response (heart rate) during the 3 minutes sit-to-stand test
Functional response during the 3 minutes sit-to-stand test: symptoms | 2 days
  Evaluate the reproductibility of functional response (symptoms) during the 3 minutes sit-to-stand test
3 minutes sit-to-stand test compared to the 6 minutes walk test: heart rate | 2 days
  Compared heart rate during the 3 minutes sit-to-stand test to the 6 minutes walk test
3 minutes sit-to-stand test compared to the 6 minutes walk test: symptoms | 2 days
  Compared symptoms during the 3 minutes sit-to-stand test to the 6 minutes walk test
1 minute sit-to-stand test compared to 3 minutes sit-to-stand: heart rate | 2 days
  Compared heart rate during the 3 minutes sit-to-stand test with 1 minute sit-to-stand test
1 minute sit-to-stand test compared to 3 minutes sit-to-stand: symptoms | 2 days
  Compared symptoms during the 3 minutes sit-to-stand test with 1 minute sit-to-stand test

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Grenoble Alpes, La Tronche
  - Groupement Hospitalier Est, Lyon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] King TE Jr, Pardo A, Selman M. Idiopathic pulmonary fibrosis. Lancet. 2011 Dec 3;378(9807):1949-61. doi: 10.1016/S0140-6736(11)60052-4. Epub 2011 Jun 28. PMID 21719092
- [Result] Cottin V, Crestani B, Valeyre D, Wallaert B, Cadranel J, Dalphin JC, Delaval P, Israel-Biet D, Kessler R, Reynaud-Gaubert M, Cordier JF, Aguilaniu B, Bouquillon B, Carre P, Danel C, Faivre JB, Ferreti G, Just N, Kouzan S, Lebargy F, Marchand Adam S, Philippe B, Prevot G, Stach B, Thivolet-Bejui F; French National Reference and Competence Centers for Rare Diseases; Societe de Pneumologies de Langue Francaise. [French practical guidelines for the diagnosis and management of idiopathic pulmonary fibrosis. From the National Reference and the Competence centers for rare diseases and the Societe de Pneumologie de Langue Francaise]. Rev Mal Respir. 2013 Dec;30(10):879-902. doi: 10.1016/j.rmr.2013.09.007. Epub 2013 Oct 25. No abstract available. French. PMID 24314711
- [Result] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Result] Nalysnyk L, Cid-Ruzafa J, Rotella P, Esser D. Incidence and prevalence of idiopathic pulmonary fibrosis: review of the literature. Eur Respir Rev. 2012 Dec 1;21(126):355-61. doi: 10.1183/09059180.00002512. PMID 23204124
- [Result] Huang XF, Gao F, Xue ZQ, Wang Y, Xu GW. [Multifactorial analysis of survival in breast cancer]. Zhonghua Zhong Liu Za Zhi. 1988 Mar;10(2):117-9. Chinese. PMID 3208648
- [Result] du Bois RM, Weycker D, Albera C, Bradford WZ, Costabel U, Kartashov A, Lancaster L, Noble PW, Sahn SA, Szwarcberg J, Thomeer M, Valeyre D, King TE Jr. Six-minute-walk test in idiopathic pulmonary fibrosis: test validation and minimal clinically important difference. Am J Respir Crit Care Med. 2011 May 1;183(9):1231-7. doi: 10.1164/rccm.201007-1179OC. Epub 2010 Dec 3. PMID 21131468
- [Result] Nathan SD, du Bois RM, Albera C, Bradford WZ, Costabel U, Kartashov A, Noble PW, Sahn SA, Valeyre D, Weycker D, King TE Jr. Validation of test performance characteristics and minimal clinically important difference of the 6-minute walk test in patients with idiopathic pulmonary fibrosis. Respir Med. 2015 Jul;109(7):914-22. doi: 10.1016/j.rmed.2015.04.008. Epub 2015 Apr 24. PMID 25956020
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Result] Buatois S, Miljkovic D, Manckoundia P, Gueguen R, Miget P, Vancon G, Perrin P, Benetos A. Five times sit to stand test is a predictor of recurrent falls in healthy community-living subjects aged 65 and older. J Am Geriatr Soc. 2008 Aug;56(8):1575-7. doi: 10.1111/j.1532-5415.2008.01777.x. No abstract available. PMID 18808608
- [Result] Macfarlane DJ, Chou KL, Cheng YH, Chi I. Validity and normative data for thirty-second chair stand test in elderly community-dwelling Hong Kong Chinese. Am J Hum Biol. 2006 May-Jun;18(3):418-21. doi: 10.1002/ajhb.20503. PMID 16634026
- [Result] Hill CJ, Denehy L, Holland AE, McDonald CF. Measurement of functional activity in chronic obstructive pulmonary disease: the grocery shelving task. J Cardiopulm Rehabil Prev. 2008 Nov-Dec;28(6):402-9. doi: 10.1097/HCR.0b013e31818c3c65. PMID 19008696
- [Result] Perrault H, Baril J, Henophy S, Rycroft A, Bourbeau J, Maltais F. Paced-walk and step tests to assess exertional dyspnea in COPD. COPD. 2009 Oct;6(5):330-9. doi: 10.1080/15412550903156317. PMID 19863362
- [Result] Brodin E, Ljungman S, Sunnerhagen KS. Rising from a chair: a simple screening test for physical function in predialysis patients. Scand J Urol Nephrol. 2008;42(3):293-300. doi: 10.1080/00365590701797556. PMID 18432536
- [Result] Ozalevli S, Ozden A, Itil O, Akkoclu A. Comparison of the Sit-to-Stand Test with 6 min walk test in patients with chronic obstructive pulmonary disease. Respir Med. 2007 Feb;101(2):286-93. doi: 10.1016/j.rmed.2006.05.007. Epub 2006 Jun 27. PMID 16806873
- [Result] Craig CP, Reynolds SL, Airhart JW, Staab EV. Alterations in immune responses by attenuated Venezuelan equine encephalitis vaccine. I. Adjuvant effect of VEE virus infection in guinea pigs. J Immunol. 1969 May;102(5):1220-7. No abstract available. PMID 4181548
- [Result] Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID 10501650
- [Result] Passing H, Bablok. A new biometrical procedure for testing the equality of measurements from two different analytical methods. Application of linear regression procedures for method comparison studies in clinical chemistry, Part I. J Clin Chem Clin Biochem. 1983 Nov;21(11):709-20. doi: 10.1515/cclm.1983.21.11.709. PMID 6655447
- [Result] Carstensen B. Comparing methods of measurement: Extending the LoA by regression. Stat Med. 2010 Feb 10;29(3):401-10. doi: 10.1002/sim.3769. PMID 19998394